CLINICAL TRIAL: NCT03596697
Title: A Randomized, Partially-blinded, Placebo-controlled, Ascending Sequential Dose Groups, Single Dose Study of the Safety, Tolerability and Pharmacokinetics of CRV431, Alone and In Combination With Tenofovir Disoproxil Fumarate in Healthy Subjects, With a Pilot Study of Multiple Ascending Sequential Doses in Healthy Volunteer Subjects
Brief Title: A Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hepion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTRV-CRV431-101
Record Dates: First submitted 2018-07-03; First posted 2018-07-24 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis B; Infectious Disease; Liver Diseases
Keywords: CRV431; Hepatitis B Virus; Hepatitis Virus
MeSH Terms: conditions — Hepatitis B; Communicable Diseases; Liver Diseases | interventions — CRV-431

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CRV431 (Experimental): Either single or multiple doses of varying dose levels
  Interventions: Drug: CRV431
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TDF (Experimental): 300 mg TDF
  Interventions: Drug: TDF

INTERVENTIONS:
Drug: CRV431 — Single or multiple dose(s) of CRV431
  Arms: CRV431
Drug: Placebo — Single Placebo dose
  Arms: Placebo
Drug: TDF — Single or multiple dose(s) of TDF
  Arms: TDF

SUMMARY:
This is three part study that will, in part one assess the safety, tolerability, and PK of a single dose of CRV431 in healthy volunteers. The second part of the study will be a single dose drug-drug interaction study in healthy volunteers with CRV431 co-treated with TDF. The third part of the study will assess the safety, tolerability, PK, and preliminary signal for antiviral efficacy and identification of clinically-relevant biomarkers of CRV431 with TDF in stable HBV patients.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent
* Willing and able to complete all study requirements
* Healthy male or female between 18 and 55 years of age (inclusive);
* Body mass index 16 to 32 kg/m2 (inclusive);

Exclusion Criteria:

* Positive test for HCVAb or HIVAb. For healthy subjects only: positive test for HBsAg
* Current or history of abuse of alcohol or illicit drugs
* Received an investigational drug, vaccine or medical device within 90 days prior to first dose of study drug.

Additional Exclusion Criteria for HBV Pilot Subjects Only:

* Evidence of significant liver fibrosis or cirrhosis
* History of NAFLD or NASH
* Positive test for HDV

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Number of healthy volunteers and patients with chronic HBV infection with treatment-related adverse events | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Jill Greytok, Study Director — ContraVir Pharmaceutical, Inc.
Locations (3):
- United States (3):
  - Celerion, Inc, Tempe, Arizona
  - Celerion, Inc, Lincoln, Nebraska
  - Pinnacle Clinical Research, San Antonio, Texas